CLINICAL TRIAL: NCT02361567
Title: Comparison of Tramacet Versus Percocet in Post Surgical Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 103278
Record Dates: First submitted 2015-02-06; First posted 2015-02-11 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Post Operative Pain
Keywords: Post Operative Pain; Addiction
MeSH Terms: conditions — Pain, Postoperative; Behavior, Addictive | interventions — Tramadol; Acetaminophen; oxycodone-acetaminophen; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tramacet (Active Comparator): Tramacet 1-2 tabs PO q4h prn
  Interventions: Drug: Tramacet
- Percocet (Active Comparator): Percocet (5/325) 1-2 tab PO q4h PRN
  Interventions: Drug: Percocet

INTERVENTIONS:
Drug: Tramacet — Pain medication commonly used post-operatively
  Other Names: tramadol/acetominophen
  Arms: Tramacet
Drug: Percocet — Pain medication commonly used post-operatively
  Other Names: oxycodone/acetominophen
  Arms: Percocet

SUMMARY:
Opioid naive patients are randomized to receive either TRAMACET or PERCOCET at the time of discharge following mild to moderate pain risk surgery. The following will be assessed: 1) Brief pain inventory (BPI) for the month. 2) Post operative pain management satisfaction. 3) Whether they sought any repeat opioid prescription. 4) Whether they intend to seek repeat opioid prescription. It is expected that both groups will have similar pain outcomes but those patients in the Percocet group will be more likely to seek a second prescription.

DETAILED DESCRIPTION:
Patient operating lists will be screened on a daily basis at identify potential patient candidates. The surgeon of note will be consulted to ensure that each patient, in their opinion, may be a candidate. If approved by the surgeon of note, the patient will then be approached in the preoperative area by a member of the research team to determine if they will consent to enrollment in the study.

Patients will be double blinded and randomized following low to moderate pain surgery (surgery in which patients do not generally require a patient controlled analgesic pump post-operatively, or require post operative analgesia beyond 14 days) to receive either tramacet 1-2 tablets orally every 4 hours prn or percocet 1-2 tablets orally every 4 prn. At time of discharge patients will recieve unidentifiable tablets in an unidentifying container of the usual dispense amount that their surgeon would standardly prescribe(range is usually between 30 and 60 tabs).

At 6 weeks patients will receive a phone call to determine a) brief pain inventory score for the month. B) if they sought a second opioid prescription. C) if they plan to seek a second script. E) satisfaction of post operative pain control on a 1-10 numerical scale f) any adverse side effects.

ELIGIBILITY:
Inclusion Criteria age 18-65

opioid naïve

postoperative from mild to moderate pain risk surgery (surgery in which patients do not generally require a patient controlled Analgesic pump post-operatively, or require post operative analgesia beyond 14 days)

Exclusion Criteria:

Patients on Opioids

Children < 18 years

Elderly

Pregnancy

Language barrier

Past medical history of psychosis

Coexisting use of anti-depressants

American Society of Anesthesia Risk Score >3

Known allergy to opioid or acetaminophen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Sought Second Prescription | 6 weeks post-operative
  What patients have sought a second opioid prescription post operatively

CONTACTS AND LOCATIONS:
Overall Officials: Collin Clarke, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- Victoria Hospital, London, Ontario, Canada